CLINICAL TRIAL: NCT01065194
Title: Efficacy and Safety of Pulsed Infusions of Levosimendan in Outpatients With Advanced Heart Failure - A Multicenter, Double-blind, Placebo Controlled Prospective Trial With Two Arms
Brief Title: Efficacy and Safety of Pulsed Infusions of Levosimendan in Outpatients With Advanced Heart Failure
Acronym: LevoRep
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Medical University Innsbruck, Department of Internal Medicine III / Cardiology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-007407-86
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2009-08

CONDITIONS: Chronic Stable Heart Failure
MeSH Terms: interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levosimendan (Experimental): Chronic stable heart failure
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator): Chronic Stable Heart Failure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levosimendan — Levosimendan will be infused on an outpatient basis for six hours at a dosage of 0,2 μg/kg/min without a bolus
  Arms: Levosimendan
Drug: Placebo — Levosimendan will be infused on an outpatient basis for six hours at a dosage of 0,2 μg/kg/min without a bolus.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effects of a pulsed application of Levosimendan versus placebo on the composite end-point functional capacity and quality of life.

DETAILED DESCRIPTION:
BACKGROUND Significant advances have been made in the treatment of congestive heart failure (CHF) in the past few years. Neurohumoral therapy with ACE-inhibitors, ß-blockers and aldosterone antagonists has been established to significantly reduce morbidity and mortality. However, despite the advances of modern therapy advanced CHF remains a syndrome with a poor prognosis. Additionally, this syndrome is associated with poor quality of life and leads to progressive debiliation and cardial cachexia. Repeat hospitalizations for acute heart failure are common among severe CHF patients. Besides the discomfort for the patients hospital admissions constitute the lion's share of the health expenditure for the heart failure syndrome.

Inotropic support is provided to patients suffering acute heart failure refractory to neurohumoral therapy. This approach is performed according to the AHA/ACC- as well as to ESC Guidelines for therapy of CHF. Inotropic therapy is targeted on hemodynamic stabilization, improvement of functional status, and reduction of rehospitalization.

Moreover, in many centres treatment with inotropes such as dobutamine and milrinone are an integral part of the applied bridge to transplant concept in severe heart failure patients. In fact, continuous or pulsed inotropic support in severe heart failure patients has been tested repeatedly in small clinical studies.

Intermittent ambulatory low dose administration of dobutamine versus conventional therapy did not improve functional capacity in the DICE-Trial. By contrast, several case series with different dose regimens of dobutamine indicated improvement of functional status.

TRIAL RATIONALE Based on its pharmacologic profile Levosimendan appears to be promising in the treatment of severe chronic heart failure functional NYHA class III/IV to improve quality of life and physical activity and to reduce hospital admissions for acute heart failure.

Repeat drug administration may be superior over a single shot therapy to maintain beneficial long-term results.

For economical reasons and for the sake of the patients comfort drug administration should ideally be managed on an outpatient basis rather than in the hospital. Therefore and for practical reasons, a time period of six hours for drug administration might be reasonable.

Dosing of the drug will be based on the experiences in the Russlan Trial and on a small case report by Martys. In the latter study serial administration of levosimendan for 6 hours (bolus of 12 mcg/kg followed by a continuous infusion of 0,1 μg/kg/min for 50min and 0,2 μg/kg/min for the next 5 hours) induced a significant fall of BNP.

In an outpatient setting, however, a bolus should be not be given for safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic stable heart failure NYHA III and IV diagnosed at least 3 months before inclusion
* 6-min.-walk-test < 350 meters
* EF < 35 %
* Age > 20 years
* Optimized and individualised neurohormonal background therapy according to ESC-guidelines for the treatment of chronic heart failure.
* Patient has signed informed consent

Exclusion Criteria:

* Hospitalization for decompensated heart failure requiring i.v. diuretics within the last month before randomization
* History of torsades des pointes
* Allergy to Levosimendan or any of the excipients
* Administration of inotropes in the last 4 weeks
* Potassium <3,5 and >5,5 mmol/l
* Systolic blood pressure <= 100 mmHg
* Women at childbearing age without using effective contraceptives ( oral contraceptives, intrauterine contraceptive devices) unless surgical sterilisation has been undertaken.
* Female patients who are pregnant or nursing
* Creatinin Clearance < 30ml/min/m2
* Severe anemia (Hb < 10 mg /dl)
* Mechanical obstruction affecting the ventricular filling or the outflow or both
* Patients with non compliance
* Severe conditions, which make the patient unsuitable to participate in a study as judged by the investigator
* Severe liver disease
* Percutaneous coronary intervention within the last 1 months
* Coronary bypass surgery within the last 3 months
* Planned HTX within the next six months
* Patient involved in another clinical trial
* De-nove heart failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
proportion of patients showing an improvement in the six-minutes walk test and a higher scoring in the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 24 weeks

SECONDARY OUTCOMES:
effects of a pulsed application of levosimendan on event free survival | 8 weeks from randomization
effects of a pulsed application of levosimendan on event free survival | 24 weeks from randomization

CONTACTS AND LOCATIONS:
Overall Officials: Johann Altenberger, MD, Principal Investigator — Paracelsus Medical University
Locations (11):
- Austria (8):
  - Medical University Innsbruck, Innsbruck
  - Allg. öffentliches Krankenhaus der Elisabethinen, Linz
  - Krankenhaus der Barmherzigen Schwestern, Linz
  - Allgemeine Krankenhaus der Stadt Linz, Linz
  - Paracelsus Medical University Salzburg, Salzburg
  - Landesklinikum St. Poelten, Sankt Pölten
  - Kaiserin Elisabeth Spital Vienna, Vienna
  - Klinikum Wels Grieskirchen, Wels
- Greece (3):
  - G. Gennimatas General Hospital, Athens
  - Hippokration General Hospital, Athens
  - Heart Failure Clinic, Attikon University Hospital, Athens

REFERENCES:
- [Derived] Altenberger J, Parissis JT, Costard-Jaeckle A, Winter A, Ebner C, Karavidas A, Sihorsch K, Avgeropoulou E, Weber T, Dimopoulos L, Ulmer H, Poelzl G. Efficacy and safety of the pulsed infusions of levosimendan in outpatients with advanced heart failure (LevoRep) study: a multicentre randomized trial. Eur J Heart Fail. 2014 Aug;16(8):898-906. doi: 10.1002/ejhf.118. Epub 2014 Jun 11. PMID 24920349